CLINICAL TRIAL: NCT05783635
Title: Reducing Alcohol Use Among Elective Surgical Patients Using Adaptive Interventions
Brief Title: Alcohol Screening and Preoperative Intervention Research Study - 2
Acronym: ASPIRE-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Anne Fernandez, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00208317; R01AA029666 (NIH)
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Drinking
Keywords: Surgery
MeSH Terms: conditions — Alcohol Drinking | interventions — Postoperative Period

STUDY DESIGN:
Intervention Model Description: The proposed study will achieve this using a Sequential Multiple Assignment Randomized Trial (SMART) design.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Enhanced Usual Care then Usual Surgical Care (Experimental): Randomized two times (2 possible randomization groups each time). Responder to Enhanced Usual Care
  Interventions: Behavioral: Enhanced Usual Care (pre-operative); Behavioral: Usual surgical care (post-operative)
- Enhanced Usual Care then Post-operative Health Coaching (Experimental): Randomized two times (2 possible randomization groups each time). Responder to Enhanced Usual Care
  Interventions: Behavioral: Enhanced Usual Care (pre-operative); Behavioral: Postoperative Virtual Health Coaching
- Enhanced Usual Care then On-Track (Experimental): Randomized two times (2 possible randomization groups each time). Non-responder to Enhanced Usual Care
  Interventions: Behavioral: Enhanced Usual Care (pre-operative); Behavioral: On-Track (Post-operative)
- Enhanced Usual Care then Combine (Postoperative Health Coaching + On-track) (Experimental): Randomized two times (2 possible randomization groups each time). Non-responder to Enhanced Usual Care
  Interventions: Behavioral: Enhanced Usual Care (pre-operative); Behavioral: Postoperative Virtual Health Coaching; Behavioral: On-Track (Post-operative)
- Enhanced Usual Care alone (Other): Only completed first randomization. Study withdrawal prior to re-randomization
  Interventions: Behavioral: Enhanced Usual Care (pre-operative)
- Preoperative Virtual Health Coaching then Usual Surgical Care (Experimental): Randomized two times (2 possible randomization groups each time). Responder to Preoperative Virtual Health Coaching
  Interventions: Behavioral: Preoperative Virtual Health Coaching; Behavioral: Usual surgical care (post-operative)
- Preoperative Virtual Health Coaching then Postoperative Virtual Health Coaching (Experimental): Randomized two times (2 possible randomization groups each time). Responder to Preoperative Virtual Health Coaching
  Interventions: Behavioral: Preoperative Virtual Health Coaching; Behavioral: Postoperative Virtual Health Coaching
- Preoperative Virtual Health Coaching then On-Track (Experimental): Randomized two times (2 possible randomization groups each time). Non-responder to Preoperative Virtual Health Coaching
  Interventions: Behavioral: Preoperative Virtual Health Coaching; Behavioral: On-Track (Post-operative)
- Preoperative Virtual Health Coaching then Combine (Postoperative Virtual Health Coaching + On-track) (Experimental): Randomized two times (2 possible randomization groups each time). Non-responder to Preoperative Virtual Health Coaching
  Interventions: Behavioral: Preoperative Virtual Health Coaching; Behavioral: Postoperative Virtual Health Coaching; Behavioral: On-Track (Post-operative)
- Preoperative Virtual Health Coaching only (Other): Only completed first randomization. Study withdrawal prior to re-randomization.
  Interventions: Behavioral: Preoperative Virtual Health Coaching

INTERVENTIONS:
Behavioral: Enhanced Usual Care (pre-operative) — The enhanced usual care will receive standard surgical care, and a resource brochure including basic information on health, alcohol use withdrawal risks, and treatment/emergency resources. The resource brochure will be e-mailed to patients or sent via postal mail.
  Arms: Enhanced Usual Care alone; Enhanced Usual Care then Combine (Postoperative Health Coaching + On-track); Enhanced Usual Care then On-Track; Enhanced Usual Care then Post-operative Health Coaching; Enhanced Usual Care then Usual Surgical Care
Behavioral: Preoperative Virtual Health Coaching — Preoperative Virtual Coaching is based on principles of health coaching, collaborative care, and motivational interviewing. Health and educational content is framed using the Health Belief Model. During two sessions, that take place approximately 3 and 5 weeks prior to surgery, the health coach presents alcohol use reduction/abstinence as important for surgical health (rather than addiction or chronic health reasons) and engages participants in discussion and patient-centered goal-setting.
  Participants will also receive a brochure including basic information on health, alcohol use withdrawal risks, and treatment/emergency resources.
  Arms: Preoperative Virtual Health Coaching only; Preoperative Virtual Health Coaching then Combine (Postoperative Virtual Health Coaching + On-track); Preoperative Virtual Health Coaching then On-Track; Preoperative Virtual Health Coaching then Postoperative Virtual Health Coaching; Preoperative Virtual Health Coaching then Usual Surgical Care
Behavioral: Usual surgical care (post-operative) — This group will receive standard post-operative care.
  Arms: Enhanced Usual Care then Usual Surgical Care; Preoperative Virtual Health Coaching then Usual Surgical Care
Behavioral: Postoperative Virtual Health Coaching — Postoperative Virtual Coaching uses the same framework and structure as Preoperative Virtual Coaching. These sessions will be delivered by a health coach using a collaborative, and motivational interviewing-based approach. The goal of these sessions is to promote well-being and help participants maintain alcohol abstinence or reduction long-term (or initiate change in alcohol use if they have not already). These sessions promote low-risk alcohol use, provide education on chronic health effects of heavy alcohol use, and teach skills for coping with or avoiding triggers for alcohol use including coping with stress and mood challenges. These sessions introduce skills to help participants manage alcohol, stress, and mood as they recover from surgery.
  Arms: Enhanced Usual Care then Combine (Postoperative Health Coaching + On-track); Enhanced Usual Care then Post-operative Health Coaching; Preoperative Virtual Health Coaching then Combine (Postoperative Virtual Health Coaching + On-track); Preoperative Virtual Health Coaching then Postoperative Virtual Health Coaching
Behavioral: On-Track (Post-operative) — On-Track is a mobile and web-accessible health tool that uses self-monitoring and provision of feedback on progress towards goals to engage participants in self-management of alcohol use and motivate behavior change through increased self-awareness and accountability for health.
  The On-Track application includes a) daily tracking of alcohol and other substance use; b) daily tracking of stress, mood, and pain; c) personalized health goals; and d) visual displays of alcohol use, stress, mood, pain, and goal achievement including graphs of trends over time.
  On-Track also uses novel monetary and non-monetary incentives to encourage utilization including an escalating monetary incentive schedule for self-monitoring.
  Arms: Enhanced Usual Care then Combine (Postoperative Health Coaching + On-track); Enhanced Usual Care then On-Track; Preoperative Virtual Health Coaching then Combine (Postoperative Virtual Health Coaching + On-track); Preoperative Virtual Health Coaching then On-Track

SUMMARY:
This sequential, multiple assignment, randomized trial will test treatments designed to reduce alcohol use before and after surgery to promote surgical health and long-term wellness.

ELIGIBILITY:
Inclusion Criteria:

1. Completed consent form, baseline survey, and enrollment phone call
2. Willingness to comply with all study procedures and availability for the duration of the study
3. Scheduled for select major elective surgery (non-cancer) in the next 5-12 weeks
4. Score ≥ 5 on the Alcohol Use Disorders Identification Test-Concise (AUDIT-C) based on research linking this score with increased risk of surgical complications
5. Access to a smart device or computer access with internet or wi-fi connection throughout the study period

Exclusion Criteria:

1. Exclude participants enrolled in another research study focused on alcohol use
2. History of severe alcohol withdrawal
3. Unable to speak, understand, or read English

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption as measured by the timeline follow-back | 10 months after surgical discharge
  Alcohol consumption will be assessed using the 30-day Timeline Follow-Back (TLFB). The TLFB will capture information on the frequency and quantity of alcohol use including average drinks/day.

SECONDARY OUTCOMES:
World Health Organization Drinking (WHO) Risk Level | 10 months after surgical discharge
  WHO drinking risk levels derived from patient reports of the number of standard drinks (defined as 0.6 ounces of absolute alcohol) consumed, converted to grams of pure alcohol (0.6 ounces = 14 grams). Ranging from abstinence (0 grams) to very high risk (101+ males / 61+ females grams).
Alcohol Use Disorder Identification test (AUDIT) | Up to 10 months after surgical discharge
  We will calculate participant's total score on the AUDIT measure. Scores on the AUDIT range from 0 to 40 with higher numbers indicating greater problematic alcohol use and presence of more alcohol use disorder symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Fernandez, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
National Institute on Alcohol Abuse and Alcoholism (NIAAA)-funded investigators conducting applicable human subjects research are expected to submit de-identified, individual-level data to this data archive. The data generated in this grant will also be presented at national or international meetings (e.g., Research Society on Alcoholism, Addiction Health Services Research, etc.) and published in a timely fashion. All final peer-reviewed manuscripts that arise from this proposal will be submitted to the digital archive in PubMed Central.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The research team will share data with NIAAA data archive (NIAAADA) biannually per funder requirements. The data in the NIAAADA are catalogued and made available to the general research community at the time of an associated publication or end of the award/support period, whichever comes first. Data in the NIAAADA is available indefinitely.
Access Criteria: Community of scientists interested in the study of alcohol use and related interventions. Additionally, data submitted to National Institute on Alcohol Abuse and Alcoholism Data Archive (NIAAADA) will be accessible by the general research community via NIAAADA.
URL: https://nda.nih.gov/niaaa